CLINICAL TRIAL: NCT00729625
Title: Air Muscle and Task Practice in Upper Limb Stroke Rehab
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Avery Gottfried, Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R21HD045514 (NIH); 7R21HD045514-03 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2005-04

CONDITIONS: Stroke
Keywords: stroke, rehabilitation, robotics
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: robotic device — The device has a small "air muscle" that when activated will slowly lift their fingers and wrist from your resting wrist position. This device is classified as a non-significant risk device by the FDA (see attached letter dated 1-15-05). The patient should not experience any pain or discomfort during this stretching activity. If they do experience any pain or discomfort they can activate a stop switch located on the control box with their unimpaired hand.
  Other Names: KMI Hand Mentor

SUMMARY:
Many patients who have sustained strokes are unable to effectively use their hemiparetic upper extremity. Limited mobility in the performance of daily activities, such as eating or dressing, adversely affects their quality of life and compromises independence. Rehabilitation techniques engaging the hemiparetic limb in repetitive task practice (RTP) may improve upper extremity function and quality of life in patients with stroke, but costs limit the number of patients that can utilize this type of therapy. Advances in microprocessor design and function make the use of an assistive device as an adjunct to RTP plausible. An innovative assistive repetitive motion (ARM) device using an "air muscle" has been developed specifically for the rehabilitation of the hemiparetic upper extremity. The primary aim of the proposed study is to collect pilot data to estimate the clinical effectiveness of using the ARM device in conjunction with RTP to improve upper extremity motor function and the quality of life of patients with stroke. Twenty sub-acute (3 to 9 mos. post-stoke) patients will be randomized to a RTP only or ARM + RTP group. The RTP group will receive 15 days (4 hours per day) of intensive one-on-one RTP therapy. The ARM + RTP group will use the ARM device for 2 hours per day and receive 2 hours of intensive RTP per day for 15 days. Clinical motor function and quality of life measures will be taken before and after the interventions and two months later. We hypothesize that the ARM + RTP group will exhibit greater improvements in motor function and quality of life measures than the RTP only group.

DETAILED DESCRIPTION:
Specific Aim 1: Estimate the effectiveness of using an assistive repetitive motion device (ARM) in conjunction with repetitive task practice (RTP) on motor recovery of patients with sub-acute stroke. This aim will be examined by comparing pre-intervention motor performance levels with the immediate post-intervention and two months post-intervention. The primary outcome variables will be scores on the Fugl-Meyer Motor Assessment Test (FMA) and Wolf Motor Function Test (WMFT). We hypothesize patients in the RTP + ARM group will exhibit greater gains in upper extremity motor recovery/performance than the RTP and ARM only groups.

Specific Aim 2: Estimate the effectiveness of using the ARM device in conjunction with RTP on health related quality of life of patients with sub-acute stoke. This aim will be examined through the administration of clinical quality of life questionnaires. The primary outcome variable to assess health related quality of life will be change scores on the Stroke Impact Scale (SIS), controlling for depressed mood as measured by the Center for Epidemiologic Studies Depression (CES-D) scale, from the pre-, immediate post and two-month post intervention testing sessions. We hypothesize patients in the RTP + ARM group will exhibit greater improvements on quality of life measures at the two-month follow-up session than the RTP and ARM only groups.

Study Design, Methods and Procedures:

Patients will be randomized to one of the following three interventional groups: repetitive task practice, assistive repetitive motion and repetitive task practice plus assistive repetitive motion. Details regarding the activities each group will perform are below.

1. Repetitive task practice (RTP) procedure: patients in the RTP group will work closely with rehabilitation professional (supervisor) for four hours per day for three weeks. We are currently accepting applications for this position. At minimum, this individual will be a licensed Physical or Occupational Therapist with clinical experience and a desire to participate and follow the outlined research protocol.

   Patients will report to the Mellon Center at the Cleveland Clinic Foundation (CCF) around 8:00 AM each day and leave around 12:00 PM. During their stay at the CCF they will be asked to engage in a series of activities that are planned for them to use their weaker or more impaired hand and arm. We will be making some additional measures about the speed at which they can do functional activities (such as reaching and folding a towel) during the testing days immediately before and after the training period and two months after completion of the training (e.g. Wolf Motor Function Test (WMFT) and Fugl-Meyer Motor Assessment (FMA)). Quality of life will be assessed with the Stroke Impact Scale (SIS) controlling for depression using the Center for Epidemiologic Studies Depression (CES-D) scale. These clinical tests require approximately 1.5 hours to administer. Participants will also be encouraged to use their weaker hand and arm at home and during the weekends.
2. Assistive repetitive motion (ARM) procedure: Patients will report to the Mellon Center at the Cleveland Clinic Foundation (CCF) around 8:00 AM each day and leave around 12:00 PM. During their stay at the CCF they will be asked to wear an assistive device on their more impaired or affected upper extremity. This device will be placed snugly on their arm and wrist. The device has a small "air muscle" that when activated will slowly lift their fingers and wrist from your resting wrist position. This device is classified as a non-significant risk device by the FDA (see attached letter dated 1-15-05). The patient should not experience any pain or discomfort during this stretching activity. If they do experience any pain or discomfort they can activate a stop switch located on the control box with their unimpaired hand. The SIS, CES-D WMFT and FMA will be administered immediately before and after the training period and two months after completion of the training.
3. RTP + ARM Procedure: Patients will report to the Mellon Center at the Cleveland Clinic Foundation (CCF) around 8:00 AM each day and leave around 12:00 PM. During their stay at the CCF they will be asked to wear an assistive device on their more impaired or affected upper extremity for two hours. This device will be placed snugly on their arm and wrist. The device has a small "air muscle" that when activated will slowly lift the fingers and wrist from a resting wrist position. They should not experience any pain or discomfort during this stretching activity. If they experience any pain or discomfort they can activate a stop switch located on the control box with the unimpaired hand. After completion of the two hour ARM intervention they will participate in two hours of RTP therapy. During this time they will engage in a series of activities that are planned for them to use the weaker or more impaired hand and arm. The SIS, CES-D WMFT and FMA will be administered immediately before and after the training period and two months after completion of the training.

The results from this project will provide valuable data as a pre-requisite for submission of a multi-year R01 randomized clinical trial to determine the clinical efficacy of using an assistive device, such as the ARM, as an adjunct to RTP. This project has the potential to increase the availability of effective rehabilitation techniques to patients with stroke.

Inclusion criteria Patients will not be excluded because of somatosensory deficits or the nature of previous physical interventions. We will not randomize patients on the basis of side of stroke or hand dominance but will undertake secondary data analyses examining these variables. In past applications of one form of RTP, CI therapy, to chronic stroke patients in the laboratories of Taub and Miltner, there were no significant differences in treatment effects for patients with right and left-sided strokes. In previous evaluations of CI therapy, Taub did not find any difference in outcomes among the small percentage of patients with pre-morbid left dominance. Therefore, there is no reason to exclude these patients from participation. We believe that the motivation to improve use of an affected pre-stroke non-dominant upper extremity is sufficiently strong to support profound improvement from treating that limb as well as from treating the dominant limb. Distributions of dominance and hand preference have been acquired from patients meeting eligibility criteria in 1998 at several sites for determining participation of sites for the EXCITE trial and side of cerebral pathology showed remarkably equal left-right distribution.

Exclusion criteria

1. a score of less than 24 on the Folstein Mini-Mental State Examination or a score of 36 or below on the Token Test of the Multilingual Aphasia Examination
2. a first stroke less than 3 months or more than 9 months prior to the initiation of therapy
3. less than 18 years old
4. clinical judgment of excessive frailty or lack of stamina (e.g., cannot attend to instructions, stay awake, engage in functional activities, etc.)
5. serious uncontrolled medical conditions
6. excessive pain in any joint of the more affected extremity that could limit ability to cooperate with the intervention, as judged by the examining clinician
7. passive range of motion less than 45 degrees for: abduction, flexion or external rotation at shoulder, or pronation of forearm; or greater than 30 degrees flexion contracture at any finger joint (patients who pass the motor criteria specified above do not tend to have the type of pain or limitation of movement that would exclude them from treatment)
8. unable to stand independently for 2 min., transfer independently to and from the toilet or perform sit-to-stand
9. current participation in other pharmacological or physical intervention studies, or have received injections of anti-spasticity drugs into upper extremity musculature within the past 3 months, or wish to have drugs injected in the foreseeable future
10. receiving any anti-spasticity drugs orally at the time of expected participation
11. received phenol injections less than 12 months prior to receiving therapy
12. contemplating a move from proximity to the treatment site in less than 1 year from the randomization date. Prospective patients who qualify but who have profound postural instability will undergo the intervention while walking with contact guarding or, when feasible, using their leg(s) and more involved arm to propel a wheelchair.

ELIGIBILITY:
Inclusion criteria Patients will not be excluded because of somatosensory deficits or the nature of previous physical interventions. We will not randomize patients on the basis of side of stroke or hand dominance but will undertake secondary data analyses examining these variables. In past applications of one form of RTP, CI therapy, to chronic stroke patients in the laboratories of Taub and Miltner, there were no significant differences in treatment effects for patients with right and left-sided strokes. In previous evaluations of CI therapy, Taub did not find any difference in outcomes among the small percentage of patients with pre-morbid left dominance. Therefore, there is no reason to exclude these patients from participation. We believe that the motivation to improve use of an affected pre-stroke non-dominant upper extremity is sufficiently strong to support profound improvement from treating that limb as well as from treating the dominant limb. Distributions of dominance and hand preference have been acquired from patients meeting eligibility criteria in 1998 at several sites for determining participation of sites for the EXCITE trial and side of cerebral pathology showed remarkably equal left-right distribution.

Exclusion criteria

1. a score of less than 24 on the Folstein Mini-Mental State Examination or a score of 36 or below on the Token Test of the Multilingual Aphasia Examination
2. a first stroke less than 3 months or more than 9 months prior to the initiation of therapy
3. less than 18 years old
4. clinical judgment of excessive frailty or lack of stamina (e.g., cannot attend to instructions, stay awake, engage in functional activities, etc.)
5. serious uncontrolled medical conditions
6. excessive pain in any joint of the more affected extremity that could limit ability to cooperate with the intervention, as judged by the examining clinician
7. passive range of motion less than 45 degrees for: abduction, flexion or external rotation at shoulder, or pronation of forearm; or greater than 30 degrees flexion contracture at any finger joint (patients who pass the motor criteria specified above do not tend to have the type of pain or limitation of movement that would exclude them from treatment)
8. unable to stand independently for 2 min., transfer independently to and from the toilet or perform sit-to-stand
9. current participation in other pharmacological or physical intervention studies, or have received injections of anti-spasticity drugs into upper extremity musculature within the past 3 months, or wish to have drugs injected in the foreseeable future
10. receiving any anti-spasticity drugs orally at the time of expected participation
11. received phenol injections less than 12 months prior to receiving therapy
12. contemplating a move from proximity to the treatment site in less than 1 year from the randomization date. Prospective patients who qualify but who have profound postural instability will undergo the intervention while walking with contact guarding or, when feasible, using their leg(s) and more involved arm to propel a wheelchair.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | 8 Weeks

REFERENCES:
- [Derived] Kutner NG, Zhang R, Butler AJ, Wolf SL, Alberts JL. Quality-of-life change associated with robotic-assisted therapy to improve hand motor function in patients with subacute stroke: a randomized clinical trial. Phys Ther. 2010 Apr;90(4):493-504. doi: 10.2522/ptj.20090160. Epub 2010 Feb 25. PMID 20185616